CLINICAL TRIAL: NCT07150052
Title: Efficacy and Safety of an Artificial Intelligence Tool for Carbohydrate Counting (Tiabete) in Children and Adults With Type 1 Diabetes Mellitus
Acronym: Tiabete
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Caroline de Gouveia Buff Passone, HEAD OF PEDIATRIC DIABETES CLINIC - PEDIATRIC ENDOCRINOLOGIST DEPARTMENT, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: USaoPauloTiabete
Record Dates: First submitted 2025-06-28; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-06

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes; technology; artificial intelligence; carb counting
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Use of Tiabete - AI tool (Experimental): Patients will use the AI tool and we will compare before and after the intervention
  Interventions: Other: Artifical intelligence in whatsapp

INTERVENTIONS:
Other: Artifical intelligence in whatsapp — AI-based tool Tia Bete, designed to assist patients with T1DM in carbohydrate counting and insulin dose adjustment. The tool provides real-time recommendations based on personalized insulin-to-carbohydrate ratios, insulin sensitivity factors, and individualized glycemic goals.

SUMMARY:
IntroductionType 1 Diabetes Mellitus (T1DM) requires lifelong exogenous insulin therapy, along with self-management strategies, such as carbohydrate counting, to appropriately adjust insulin doses in response to meals. However, many patients face challenges in adhering consistently to carbohydrate counting, compromising glycemic control and increasing the risk of diabetes-related complications. Emerging technologies, such as artificial intelligence (AI), hold significant potential for optimizing disease management by enhancing the accuracy and efficiency of self-care practices. ObjectiveThe primary aim of this study is to evaluate the efficacy and safety of the AI-based tool Tia Bete, designed to assist patients with T1DM in carbohydrate counting and insulin dose adjustment. The tool provides real-time recommendations based on personalized insulin-to-carbohydrate ratios, insulin sensitivity factors, and individualized glycemic goals. MethodsThis is a prospective, longitudinal study involving 40 patients with T1DM, stratified into two cohorts: 20 children and adolescents (6-18 years) and 20 adults (>18 years), recruited at the Hospital das Clínicas, University of São Paulo (HCFMUSP). Participants will be assessed before and after six months of using the Tia Bete tool. Glycemic control will be evaluated using parameters such as glycated hemoglobin (HbA1c), time in range, and the incidence of hypoglycemia and hyperglycemia. Quality of life and satisfaction with the tool will also be assessed. Overview of the AI Tool Launched in June 2024, Tia Bete is an AI-based digital solution designed to facilitate glycemic control and improve quality of life for patients with T1DM. By offering real-time assistance with carbohydrate counting and insulin dose recommendations, the tool aims to enhance patient autonomy while enabling flexible treatment adherence in collaboration with their multidisciplinary healthcare team. Results and ConclusionsPreliminary data indicate high engagement, with over 35,000 active users interacting with the platform at least four times per week. Initial findings suggest significant improvements in glycemic control, as well as increased confidence in carbohydrate counting and insulin dose adjustments. The dissemination of this project is crucial for advancing T1DM care, offering a scalable, accessible, and effective technological solution. Final results are expected by October 2025.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 1 diabetes mellitus
* children between 6 and 18 years old and their caregivers; and adults > 18 years old.

Glycated Hb between 7.2-10.5% in the last 6 months. Being on a basal-bolus regimen Participating in and understanding the guidelines on how to use the program to be tested in this study Agreeing to the free and informed consent form. Performing periodic monitoring at the DM outpatient clinic at HC-FMUSP

Exclusion Criteria:

* Not understanding the instructions.
* Being illiterate
* Not attending the visits proposed by the study
* Not using the tool via WhatsApp.
* Not accepting consent.
* Interacting with the tool less than 3 days a week during the study period.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Glycated hemoglobin (HbA1c) | 6 months
  Participants will be assessed before and after six months of using the Tia Bete tool. Glycemic control will be evaluated using :
  - Hb1 Ac ( as a percentage of total hemoglobin- real value)
- time in range ( percentage) - hypoglycemia (mean daily percentage of hypo- glycemia less than 70 mg/dl) - hyperglycemia(mean daily percentage of hyper- glycemia above than 180mg/dl) | 6 months
  Participants will be assessed before and after six months of using the Tia Bete tool. Glycemic control will be evaluated using :
  * time in range ( percentage)
  * hypoglycemia (mean daily percentage of hypo- glycemia less than 70 mg/dl)
  * hyperglycemia(mean daily percentage of hyper- glycemia above than 180mg/dl)

SECONDARY OUTCOMES:
Quality of life | 6 months
  Diabetes-specific health-related quality of life will be assessed with validated, age-appropriate instruments: the Pediatric Quality of Life Inventory (PedsQL) 3.0 Diabetes Module for children/adolescents (<18 years) and the Brazilian abridged version of the Diabetes Quality of Life Measure (DQOL-Brazil-8) for adults (≥18 years). Scores for both instruments range from 0 (lowest possible quality of life) to 100 (highest); higher scores indicate better quality of life.
Satisfaction with the tool | 6 months
  Participant satisfaction with the intervention will be assessed using the Satisfaction Form with the Tia Bete Tool. The instrument yields a total score from 4 (minimum possible satisfaction) to 30 (maximum possible satisfaction); higher scores indicate greater satisfaction with the tool.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cengiz E, Danne T, Ahmad T, Ayyavoo A, Beran D, Ehtisham S, Fairchild J, Jarosz-Chobot P, Ng SM, Paterson M, Codner E. ISPAD Clinical Practice Consensus Guidelines 2022: Insulin treatment in children and adolescents with diabetes. Pediatr Diabetes. 2022 Dec;23(8):1277-1296. doi: 10.1111/pedi.13442. No abstract available. PMID 36537533
- [Background] Annan SF, Higgins LA, Jelleryd E, Hannon T, Rose S, Salis S, Baptista J, Chinchilla P, Marcovecchio ML. ISPAD Clinical Practice Consensus Guidelines 2022: Nutritional management in children and adolescents with diabetes. Pediatr Diabetes. 2022 Dec;23(8):1297-1321. doi: 10.1111/pedi.13429. Epub 2022 Dec 5. No abstract available. PMID 36468223